CLINICAL TRIAL: NCT04502888
Title: Phase 1 Dose Escalation Study of the Agonist Redirected Checkpoint, SL-172154 (SIRPα-Fc-CD40L), Administered Intratumorally in Subjects With Cutaneous Squamous Cell Carcinoma or Squamous Cell Carcinoma of the Head and Neck
Brief Title: Ph1 Study of SL-172154 Administered Intratumorally in Subjects With Squamous Cell Carcinoma of the Head and Neck or Skin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Shattuck Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SL03-OHD-102
Record Dates: First submitted 2020-07-31; First posted 2020-08-06 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck
Keywords: intratumoral injection
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SL-172154 (Experimental): Intratumoral administration
  Interventions: Drug: Drug: SL-172154

INTERVENTIONS:
Drug: Drug: SL-172154 — The investigational product (IP), SL-172154, is a novel fusion protein consisting of human SIRPα and CD40L (SIRPα -Fc-CD40L) linked via a human Fc.

SUMMARY:
This is a Phase 1 open-label, multi-center, dose-escalation study to evaluate the safety, PK, anti-tumor activity, and pharmacodynamic effects of SL-172154 administered by intratumoral injection in subjects with cutaneous squamous cell carcinoma (CSCC) or squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
This Phase 1 trial will evaluate the safety, tolerability, pharmacokinetics, anti-tumor activity and pharmacodynamic effects of SL-172154 when administered as an intratumoral injection (ITI) and identify the dose and schedule i.e., recommended Phase 2 dose (RP2D) for future development. Eligible subjects must have unresectable or recurrent, locally advanced or metastatic squamous cell carcinoma of the skin or head and neck, that is not amenable to curative surgery or radiotherapy. The study design consists of four sequential dose-escalation cohorts and an optional pharmacodynamic cohort to obtain additional pharmacodynamic data at one or more dose levels that have completed evaluation for safety without exceeding the maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Subject has voluntarily agreed to participate by giving written informed consent in accordance with ICH/GCP guidelines and applicable local regulations.
* Subject must have a histologically confirmed diagnosis of an unresectable or recurrent, locally advanced or metastatic cutaneous squamous cell carcinoma or squamous cell carcinoma of the head and neck that is not amenable to curative surgery or radiotherapy.
* Subjects must have received, been intolerant to, or ineligible for standard therapy(ies) known to provide clinical benefit for their condition.
* Subject has measurable disease by RECIST v1.1 using radiologic assessment.
* Subject has at least 1 tumor lesion measuring between 1-6cm that is cutaneous and/or subcutaneous and/or nodal and is clinically accessible and safe for injection by direct visualization, palpation or by ultrasound guidance. PD Cohort Subjects Only: Must have a second lesion that is non-injected and is amenable to tumor biopsy collection.
* Subject age is 18 years and older.
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Has life expectancy of greater than 12 weeks.
* Has adequate organ function.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 72 hours of D1 of IP.
* Male subjects of reproductive potential must use acceptable contraception.
* Recovery from prior anti-cancer treatments including surgery, radiotherapy, chemotherapy or any other anti-cancer therapy to baseline or ≤ Grade 1.
* Willing to consent to mandatory pre-treatment and on-treatment tumor biopsy(ies) of injected lesion (and non-injected lesion(s) for subjects enrolled in the PD cohort)

Exclusion Criteria:

* Prior treatment with an anti-CD47 or anti-SIRPα targeting agent or a CD40 agonist.
* Any anti-cancer therapy within the washout period prior to first dose (D1) of SL-172154.
* Concurrent chemotherapy, immunotherapy, biologic or hormonal/hormonal suppression therapy for cancer treatment is prohibited. Concurrent use of hormones for non-cancer related conditions is acceptable.
* Use of corticosteroids or other immunosuppressive medication, current or within 14 days of D1 of SL-172154 treatment.
* Receipt of live attenuated vaccine within 28 days of D1 of IP.
* Hypersensitivity to the active drug substance or to any of the excipients for the agent to be administered or subjects with known hypersensitivity to Chinese hamster ovary cell products.
* History of coagulopathy resulting in uncontrolled bleeding, eg, hemophilia, von Willebrand's disease.
* Requires continuous anticoagulation therapy or antiplatelet therapy
* Active or documented history of autoimmune disease. Exceptions include controlled Type I diabetes, vitiligo, alopecia areata or hypo/hyperthyroidism.
* Active pneumonitis (i.e. drug-induced, idiopathic pulmonary fibrosis, radiation-induced, etc.).
* Ongoing or active infection (e.g., no systemic antimicrobial therapy for treatment of infection within 5 days of D1 of IP).
* Symptomatic peptic ulcer disease or gastritis, active diverticulitis, other serious gastrointestinal disease associated with diarrhea within 6 months of D1 of IP.
* Clinically significant or uncontrolled cardiac/thromboembolic disease.
* Untreated central nervous system or leptomeningeal metastases.
* Women who are breastfeeding.
* Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs or compromised ability to provide written informed consent.
* Another malignancy that requires active therapy and that in the opinion of the investigator and Sponsor would interfere with monitoring of radiologic assessments of response to IP.
* Has undergone allogeneic stem cell transplantation or organ transplantation.
* Known history or positive test for human immunodeficiency virus, or positive test for hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- SL-172154 (0.003 mg): 0.003 mg of SL-172154 via intratumoral injection
- SL-172154 (0.01 mg): 0.01 mg of SL-172154 via intratumoral injection
Period: Overall Study
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 3 | 1 | 4
Age, Continuous [Median (Full Range); unit: years] | 70.0 [67 to 82] | 63.5 [56 to 71] | 70.0 [56 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Cancer type [Number; unit: participants]
  cutaneous squamous cell carcinoma | 3 | 1 | 4
  squamous cell carcinoma of the head and neck | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All Treatment Emergent Adverse Events
Description: Number of participants with treatment-emergent adverse events
Time Frame: From Day 1 to 90 days after last injection of SL-172154, an average of 6 weeks. SL-172154 administration continued until disease progression or withdrawal of consent; there was no maximum treatment duration.
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of SL-172154 When Administered Intratumorally
Description: Number of participants with dose limiting toxicities (DLTs)
Time Frame: From Day 1 to Day 29.
Population: DLT evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

3. Secondary Outcome: Establish the Recommended Phase 2 Dose (RP2D) for SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Based on review of all data, including safety, tolerability, PK, anti-tumor activity and PD effects
Time Frame: Approximately 18-24 months
Measure: Number; unit: mg
Groups:
- SL-172154: Intratumoral SL-172154 given on Days 1, 8, and 15 of Cycle 1 (21 days) and Day 1 of all additional cycles (21 days each)
Arm/Group | SL-172154
Number analyzed (Participants) | 5
mg | NA — Study was terminated early, prior to determination of the RP2D

4. Secondary Outcome: Objective Response Rate of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Number of participants with an objective response per investigator assessment according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1). Objective response includes complete response (disappearance of all target lesions) and partial response (>/= 30% decrease in the sum of the longest diameter of target lesions).
Time Frame: Approximately 18-24 months
Population: Response Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

5. Secondary Outcome: Immunogenicity to SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Proportion of participants with positive anti-drug antibody titer
Time Frame: Approximately 18-24 months
Population: Due to the small number of subjects and limited systemic exposure SL-172154 by ITI, samples were not analyzed for the presence of anti-drug antibodies to SL-172154.
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Maximum Observed Concentration (Cmax) of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: The Cmax is the maximum observed serum concentration of SL-172154 following single and multiple doses
Time Frame: Approximately 18-24 months
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
ng/mL | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

7. Secondary Outcome: Time at Which the Maximum Concentration is Observed (Tmax) of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: The Tmax is the time at which the maximum concentration of SL-172154 is observed following single and multiple doses
Time Frame: Approximately 18-24 months
Measure: Median (Full Range); unit: hours
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
hours | NA [NA to NA] — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA [NA to NA] — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

8. Secondary Outcome: Minimum Observed Concentration (Cmin) of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: The Cmin is the minimum observed serum concentration of SL-172154 following single and multiple doses
Time Frame: Approximately 18-24 months
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
ng/mL | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

9. Secondary Outcome: Area Under the Serum Concentration Time Curve (AUC) of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: The AUC is the area under the serum concentration time curve following single and multiple doses of SL-172154
Time Frame: Approximately 18-24 months
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
hours*ng/mL | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

10. Secondary Outcome: Terminal Elimination Half-life (t1/2) of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Terminal elimination half-life (t1/2) of SL-172154
Time Frame: Approximately 18-24 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
hours | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

11. Secondary Outcome: Clearance (CL) of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Clearance of Sl-172154
Time Frame: Approximately 18-24 months
Measure: Mean (Standard Deviation); unit: liters per hours
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
liters per hours | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

12. Secondary Outcome: Volume of Distribution of SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Volume of distribtion of SL-172154
Time Frame: Approximately 18-24 months
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
liters | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study. | NA (NA) — The serum concentration of SL-172154 was below the limit of quantitation in all samples collected during the study.

13. Other Pre Specified Outcome: Changes From Baseline in Cell Counts to Assess Pharmacodynamic Biomarkers in Blood Prior to, On-treatment and Following SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Circulating immune cells such as: T cells, B cells, natural killer (NK) cells, and myeloid cells and circulating chemokine and cytokine levels
Time Frame: Approximately 18-24 months
Population: Due to the small number of subjects and Sponsor decision to pursue development of SL-172154 by IV administration, a complete set of PD samples was not analyzed or reported.
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Changes From Baseline in Cell Counts to Assess Pharmacodynamic Biomarkers in Tumor Tissue Prior to, On-treatment and Following SL-172154 When Administered by Intratumoral Injection (ITI)
Description: Presence of SL-172154 in tumor tissue, changes in T cells subsets, B cells and macrophages and assessment of SL-172154 in the tumor tissue, CD47 and CD40 expression and Programmed cell death ligand 1 (PD-L1) expression
Time Frame: Approximately 18-24 months
Population: as for outcome 13
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: To Estimate Progression-free Survival (PFS)
Description: PFS: time from first dose to progression by RECIST v1.1 or death, whichever comes first
Time Frame: Approximately 18-24 months
Measure: Median (Standard Deviation); unit: weeks
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
Number analyzed (Participants) | 3 | 2
weeks | NA (NA) — Due to the small number of subjects, PFS data was not informative. | NA (NA) — Due to the small number of subjects, PFS data was not informative.

ADVERSE EVENTS:
Time Frame: Subjects were followed continuously for all AEs starting when a subject signed the informed consent form, throughout the course of treatment, and for 90 days after the last dose of study treatment, an average of 6 weeks. SL-172154 administration continued until disease progression or withdrawal of consent; there was no maximum treatment duration.
Arm/Group | SL-172154 (0.003 mg) | SL-172154 (0.01 mg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SL-172154 (0.003 mg) (N=3) | SL-172154 (0.01 mg) (N=2)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SL-172154 (0.003 mg) (N=3) | SL-172154 (0.01 mg) (N=2)
Injection site pain (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Lymph gland infection (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site agrees not to publish any Study Results or data before the publication of results from the Overall Study. After Sponsor haspublished the results of the Overall Study, Site may publish or present results generated at Site. If Sponsor has not publishedresults of the Overall Study within 18 months of data base lock, Site may publish the results of the Study that were generated atSite. Site agrees to first submit to Sponsor the proposed publication at least 30 days prior to the submission.

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT04502888/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04502888/SAP_001.pdf